CLINICAL TRIAL: NCT03449459
Title: A Randomized, Parallel, Controlled, Exploratory Study: the Efficacy and Safety of Taking Probiotics, Inhaled Antibiotics or Combined Vaccination to Prevent Acute Exacerbation in Subjects With Moderate to Severe COPD and Decolonize Bacteria in Lower Respiratory Tract.
Brief Title: Prevention of Acute Exacerbation in Subjects With COPD by Bacterial Decolonization in Lower Respiratory Tract
Acronym: PAEAN
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other); Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B2017-197R; 2017YFC1309303 (Other Grant/Funding Number: Ministry of science and technology of China.)
Record Dates: First submitted 2018-02-12; First posted 2018-02-28 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2018-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: chronic obstructive pulmonary disease; aerosol inhaled amikacin; oral probiotics; combined influenza and pneumococcal vaccine inoculation; bacterial decolonization in lower respiratory tract
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Participants are equally assigned to four groups in parallel to accept oral probiotics, aerosol inhaled amikacin, combined vaccination or blank control for the duration of the study.
Masking Description: Although this study is unblinded, we will adopt method of allocation concealment to reduce selection bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- oral probiotics (Experimental)
  Interventions: Dietary Supplement: oral probiotics
- aerosol inhaled amikacin (Experimental)
  Interventions: Drug: aerosol inhaled amikacin
- combined vaccination (Experimental)
  Interventions: Biological: combined vaccination
- conventional therapy (blank control) (No Intervention): According to the subjects' personal characteristics and guidance of The Global Initiative for Chronic Obstructive Lung Disease(GOLD) 2017, the doctor in charge prescribes appropriate medication, including but not limited to bronchodilators, inhaled glucocorticoids and long term oxygen therapy.

INTERVENTIONS:
Dietary Supplement: oral probiotics — Culturelle™ DIGESTIVE HEALTH 30 CT(VCAP)(10 Billion Claim) which consists of 100% Lactobacillus rhamnosus GG, 1 tablet, q.d., for 3 months.
  Subjects will take conventional therapy at the same time.
  Arms: oral probiotics
Drug: aerosol inhaled amikacin — 0.4g Amikacin sulfate injection + 5ml saline, aerosol inhalation, b.i.d., 5-7 days per month, for 3 months.
  In order to observe and cope with adverse events timely, subjects will be admitted to the ward during the course of medication.
  Subjects will take conventional therapy at the same time.
  Arms: aerosol inhaled amikacin
Biological: combined vaccination — Influenza Vaccine recommended by World Health Organization(WHO) in that year and imported 23-Valent Pneumococcal Polysaccharide Vaccine approved by China Food and Drug Administration(CFDA) are vaccinated at different body sites by professional nurses.
  The interval between two vaccinations is 3-5 days to avoid the overlap of adverse events.
  Subjects will take conventional therapy at the same time.
  Arms: combined vaccination

SUMMARY:
The colonization of potential pathogenic bacteria in lower respiratory tract is thought to be accountable for acute exacerbation in subjects with moderate to severe COPD. However, there is no accepted therapy for patients with COPD to remove the colonized bacteria in lower respiratory tract. Therefore, we plan to perform a multi-center, randomized, controlled trial to study the efficacy and safety of oral probiotics, aerosol inhaled amikacin or combined vaccination to decolonize bacteria in lower respiratory tract and prevent acute exacerbation of COPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a chronic respiratory disease characterized by incomplete reversible airflow limitation, small airway obstruction and alveolar structural damage. About 3 million patients die from COPD every year around the world. The prevalence of COPD in Chinese people over the age of 40 is as high as 12 % and has risen by 50 % in the past nine years.

Acute exacerbation is the leading cause of death in patients with COPD , and accounts for a majority of expenditure of COPD management. The colonization of potential pathogenic bacteria in the lower respiratory tract is an important cause of the acute exacerbation especially in patients with moderate and severe COPD.

Some clinical studies show that aerosol inhaled antibiotics is promising in reducing acute exacerbation, but these exploratory studies have some defects so that they can't back up for the clinical application of aerosol inhaled antibiotics. Amikacin, a kind of aminoglycosides, is sensitive to the common pathogens of acute exacerbation of COPD in China. Therefore it is necessary to carry out a clinical trial to verify its efficacy and safety in pathogen decolonization and prevention of acute exacerbation.

In addition, owing to bacterial resistance and insufficient antibiotics concentration in lower respiratory tract, developing new antibacterial materials is necessary. Oral probiotics is an another way to regulate the bacterial load and inflammatory response in lower respiratory tract, which has been proven to effectively prevent acute exacerbation in cystic fibrosis and childhood asthma. Likewise, airway bacterial burden and inflammation are two main mechanisms of acute exacerbation in COPD. Hence, considering its convenience and safety of oral probiotics, we perform a trial to make clinical evaluation for it.

What's more, influenza and streptococcus pneumoniae vaccines are separately recommended for patients with COPD in the Global Initiative for Chronic Obstructive Pulmonary Disease(GOLD), but there have been no studies on the effects of combined vaccination on bacterial decolonization in lower respiratory tract or on the prevention of acute exacerbation.

Effects of these above methods on the decolonization of potential pathogenic bacteria in lower respiratory tract and the inflammatory reaction are not clear. Therefore, we plan to perform a multi-center, randomized, controlled trial to study the efficacy and safety of oral probiotics, aerosol inhaled amikacin or combined vaccination to decolonize bacteria in lower respiratory tract and prevent acute exacerbation of COPD.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed
2. Male or female adults aged 18-65 years
3. Diagnosed with COPD according to GOLD 2016 (The ratio of post-bronchodilator forced expiratory volume in 1 second (FEV1) to force vital capacity (FVC)<0.70 with the use of salbutamol 400ug)
4. Moderate to very severe airflow limitation (post-bronchodilator FEV1 < 80% of the predicted normal value)
5. A documented history of at least 2 COPD exacerbation in the previous 12 months that required treatment with systemic glucocorticoids and/or antibiotics, or at least 1 exacerbation in the previous 12 months that requires hospitalization.
6. In the stable stage of COPD

Exclusion Criteria:

1. Patients who have clinically significant and chronic hepatic, renal, cardiovascular and gastrointestinal abnormalities or malignant tumor (except for lung cancer) which could interfere with the assessment of the efficacy and safety of the study treatment
2. Patients who are in critical conditions
3. Patients who have had a COPD exacerbation that required treatment with antibiotics and/or systemic corticosteroids or an acute exacerbation of any other diseases in the 4 weeks prior to screening
4. Patients with concomitant pulmonary disease (including but not limited to bronchiectasis, interstitial lung disease, asthma)
5. Patients who are highly likely to be lost during the 3-month treatment and the 1-year follow up
6. Pregnant or nursing (lactating) women
7. Patients who have been vaccinated against influenza in the current year, or against Streptococcus pneumoniae within five years, or have vaccination contraindications
8. Patients who are allergic to amikacin or other aminoglycosides
9. Patients who have participated in any interventional clinical trials in the three months prior to screening
10. Patients with mental diseases or cognitive disorders which could interfere with treatment and follow-up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Time to the first COPD exacerbation | 15 months
  COPD exacerbation refers to deterioration of patients' daily symptoms requiring treatment with antibiotics or systemic glucocorticoid therapy.
  First COPD exacerbations starting between first dose and one day after last follow-up are included.

SECONDARY OUTCOMES:
Colonization of potential pathogenic bacteria in induced sputum | Baseline, 3 months
  Induced sputum represents the specimen from lower respiratory tract and should be processed within six hours after collection. Sputum plugs were separated from contaminating saliva by macroscopic examination using sterile forceps. Haemophilus influenzae, Streptococcus pneumoniae, Moraxella catarrhalis and Pseudomonas aeruginosa which are the top four bacteria involved in acute exacerbation of COPD are defined as potential pathogenic bacteria. Using the plate count method, when the colony number of above four bacteria is over 100 cfu/ml，we define this bacteria as colonized bacteria in lower respiratory tract.
Microbiome in induced sputum | Baseline, 3 months
  Induced sputum represents the specimen from lower respiratory tract and should be processed within six hours after collection. Sputum plugs were separated from contaminating saliva by macroscopic examination using sterile forceps and weighed. Bacterial genomic DNA was isolated from sputum plugs of the same weight using the specific kits. The 16S bacterial ribosomal RNA genes were Polymerase Chain Reaction (PCR)-amplified with the appropriate controls against reagent contamination. Amplified DNA fragments were sequenced using the specific sequencing platform. Sequencing reads were processed and analyzed by the specific algorithm and software. The composition and diversity of microbiome are represented by major taxonomic groups at both phylum and genus levels. If necessary, Quantitative PCR for 16S rRNA gene will be performed to validate the results of sequencing. By using these methos, we can detect the microbiome's composition and its shift.
Forced Expiratory Volume in 1 Second | Baseline, 3 months, 15 months
  Change from baseline. Pulmonary function assessments were performed using centralized spirometry according to international standards. FEV1 was measured after 15 minutes of inhaling salbutamol 400ug.
COPD Assessment Test(CAT) Score | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months
  The COPD Assessment Test (CAT) is an 8-item uni-dimensional measure of health status impairment in COPD, containing 6 grades from 0 to 5.
modified Medical Research Council(mMRC) scale | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months
  The modified Medical Research Council scale is a simple and powerful tool to evaluate the breathlessness, containing 5 grades from 0 to 4.
serum C-reactive protein(CRP) levels | Baseline, 3 months
  Serum CRP level is a sensitive marker of the systemic inflammation.
interleukin(IL)-6 in induced sputum | Baseline, 3 months
  Induced sputum represents the specimen from lower respiratory tract. Sputum supernatant was batch analysed for the cytokines IL-6 using commercial highsensitivity sandwich ELISA kits. Inflammatory factors represent local inflammation levels in lower respiratory tract.
IL-8 in induced sputum | Baseline, 3 months
  Induced sputum represents the specimen from lower respiratory tract. Sputum supernatant was batch analysed for the cytokines IL-8 using commercial highsensitivity sandwich ELISA kits. Inflammatory factors represent local inflammation levels in lower respiratory tract.
IL-1β in induced sputum | Baseline, 3 months
  Induced sputum represents the specimen from lower respiratory tract. Sputum supernatant was batch analysed for the cytokines IL-1β using commercial highsensitivity sandwich ELISA kits. Inflammatory factors represent local inflammation levels in lower respiratory tract.
Number of Patients With Adverse Events, Serious Adverse Events, and Death | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months
  The overall rate of adverse events reported from initiation to the last time follow-up. Some laboratory examinations, such as blood routine, hepatorenal function and electrocardiogram, are performed twice separately at baseline and completion of intervention(3 months) in order to evaluate the safety of interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zhang, MD, PhD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (3):
- China (3):
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Ruijin Hospital, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hua JL, Yang ZF, Cheng QJ, Han YP, Li ZT, Dai RR, He BF, Wu YX, Zhang J. Prevention of exacerbation in patients with moderate-to-very severe COPD with the intent to modulate respiratory microbiome: a pilot prospective, multi-center, randomized controlled trial. Front Med (Lausanne). 2024 Jan 5;10:1265544. doi: 10.3389/fmed.2023.1265544. eCollection 2023. PMID 38249987